CLINICAL TRIAL: NCT05048212
Title: A Phase II Study of Nivolumab With Ipilimumab and Cabozantinib in Patients With Untreated Renal Cell Carcinoma Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0520; NCI-2021-10708 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-02; First posted 2021-09-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Brain Metastases; Renal Cell Carcinoma
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab (Experimental): by vein every 3 weeks for 4 doses
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Cabozantinib
- Ipilimumab (Experimental): by vein over 30 minutes every 3 weeks for 4 doses
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Cabozantinib
- Cabozantinib (Experimental): tablets by mouth 1 time every day.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Nivolumab — Given by IV
Drug: Ipilimumab — Given by IV
Drug: Cabozantinib — Given by IV

SUMMARY:
A Phase II Study of Nivolumab with Ipilimumab and Cabozantinib in Patients with Untreated Renal Cell Carcinoma Brain Metastases

DETAILED DESCRIPTION:
This is a phase II study to assess the safety and efficacy of the combination of nivolumab with ipilimumab and cabozantinib in patients with untreated brain metastases from RCC until disease progression or intolerable toxicities or patient withdrawal. We will accrue a total of 40 patients. Patients will be treated with nivolumab (3mg/kg) and ipilimumab (1mg/kg) IV every 3 weeks for 4 doses and cabozantinib 40mg daily. Then patients will be treated with nivolumab 480mg IV Q 4 weeks and cabozantinib 40mg daily until progression or intolerable toxicities or patient's withdrawal. A lead-in group of 6 patients will be closely monitored for DLT. If stopping criteria (>3 patients develop DLTs) is met then, treatment will be switched to Nivolumab plus Cabozantinib omitting ipilimumab.

ELIGIBILITY:
Inclusion Criteria

1. Signed Informed Consent Form (ICF)
2. Ability and willingness to comply with the requirements of the study protocol
3. Age ≥18 years
4. Life expectancy >12 weeks
5. Asymptomatic and off steroids for at least 10 days except patients: who have mild symptoms from intracranial disease that do not affect their performance status
6. Prior therapies for extracranial metastatic renal cell carcinoma as long as it did not include anti- CTLA-4 or cabozantinib or MET inhibitors
7. Patients with histologically confirmed metastatic renal cell carcinoma and at least one measurable intracranial target lesion for which all of the following criteria are met:

   - Previously untreated or progressive after previous local therapy(limited to SRS and surgery)
   * Immediate local therapy clinically not indicated or patient is not a suitable candidate to receive immediate local therapy.
   * 5mm to 30mm, as determined by MRI with contrast.
8. Adequate hematologic and essential organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (C1D1)

   * Absolute neutrophil count (ANC) ≥1500 cells/µL
   * White blood cell (WBC) counts >2500/µ -- Lymphocyte count ≥500/µL
   * Platelet count ≥ 100,000/µL;
   * Hemoglobin ≥9.0 g/dL
   * Serum albumin≥2.8g/dl
   * Total bilirubin ≤1.5×upper limit of normal (ULN) with the following exception:

   Patients with known Gilbert disease who have serum bilirubin level ≤3×ULN may be enrolled.

   - Alanine aminotransferase (ALT) ≤ 3x upper limit of normal (ULN).
   * Aspartate aminotransferase (AST) ≤ 3x upper limit of normal (ULN).
   * Alkaline phosphatase ≤5×ULN in patients with documented bone metastases.
   * Serum creatinine ≤ 1.5x ULN or calculated creatinine clearance ≥ 40mL/min (≥ 0.675mL/sec) using the Cockcroft-Gault equation: Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
   * Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g.
9. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for at least 12 months after the last dose of Cabozantinib and Nivolumab
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 (see Appendix 5)
11. INR and aPTT ≤1.5×ULN within 7 days prior to study enrollment 12. Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.

Exclusion Criteria

1. Symptomatic brain metastases requiring immediate local interventions such as craniotomy or SRS or whole brain radiation.
2. Patients who require immediate surgical or radiotherapy interventions for extra-cranial lesions.
3. Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
4. Requiring corticosteroid dose in 10 days prior to administration of first dose of study drug with following exceptions

   - Symptomatic patients who have stable or decreasing corticosteroid use in the past 10 days may be included
5. Patients with Leptomeningeal disease.
6. Any approved anticancer therapy, including chemotherapy and hormonal therapy within 4 weeks prior to initiation of study treatment; however, the following are allowed:

   * Hormone-replacement therapy or oral contraceptives
   * Herbal therapy >1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1,Day 1)
7. Current, recent (within 3 weeks of the first infusion of this study), or planned participation in an experimental drug study.
8. AEs from prior anticancer therapy that have not resolved to Grade ≤1 except for alopecia.
9. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; >Childes A cirrhosis; fatty liver; and inherited liver disease.
10. Patients with acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma.
11. Patients who are pregnant, lactating, or breastfeeding.
12. Known hypersensitivity to recombinant human antibodies.
13. Inability to undergo MRI secondary to Metal implant and Gadolinium contrast allergy.
14. Inability to comply with study and follow-up procedures.
15. History of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome,

    Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis with the following exception:
    * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
    * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
    * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA), Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%).
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
16. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan with the following exception

    -History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
17. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
18. History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection with the following exception:

    * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
19. Active tuberculosis.
20. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
21. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1.
22. Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1 with the following exception.

    - Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
23. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study

    - Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study and at least 5 months after last dose of nivolumab.
24. Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score

    ≤ 6, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc.).
25. Life expectancy of less than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To associate if the combination of nivolumab with ipilimumab and cabozantinib produces improvesintracranial progression-free survival (PFS) in patients. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT05048212/ICF_000.pdf